CLINICAL TRIAL: NCT03306888
Title: Feasibility and Acceptability of Implementing a Clinic-based Physical Activity Coaching Intervention in People With Premanifest and Early Stage Huntington's Disease
Brief Title: Feasibility and Acceptability of Implementing a Clinic-based Physical Activity Coaching Intervention in People With Premanifest and Early Stage HD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 546845
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2018-11

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: Single arm feasibility study with 14 participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity Coaching Intervention (Experimental): The intervention will entail one face-to-face coaching session (approximately 1 hour) to be held approximately 1 week following the baseline assessment, and three remote video sessions (via secure Webex connection via computer or smart phone, or phone call if internet/smart phone is not available to participant) lasting approximately 20 minutes.
  Interventions: Other: Physical Activity Coaching

INTERVENTIONS:
Other: Physical Activity Coaching — Physical activity coaching over 4 months

SUMMARY:
This study will evaluate the feasibility and acceptability of a clinic-based physical activity coaching intervention in people with pre-manifest and early stage Huntington's Disease (HD). Fourteen individuals with premanifest and early stage HD will be recruited to participate in a 4 month coaching intervention. Feasibility will be assessed by recruitment and retention rates, and acceptability will be assessed by participant interviews. Participants will also be evaluate at baseline and following the coaching intervention to explore preliminary efficacy in terms of physical activity, self efficacy, disease-specific motor and cognitive function, walking endurance and strength.

DETAILED DESCRIPTION:
The investigators have previously developed and evaluated a physical activity behavioral change intervention in people with early-mid stage HD (Engage-HD). In a study conducted in the United Kingdom, self-reported physical activity, self-efficacy for exercise, and cognition were increased for those in the coaching intervention group compared to a social contact control group. This intervention has not yet been applied to individuals with pre-manifest (prior to onset of clinical symptoms) and early stage HD, where it may be most critical to engage in exercise. To date, no study has prospectively evaluated a physical activity intervention to facilitate exercise uptake in these earliest stages. This study will explore the feasibility and acceptability of the Engage-HD intervention in 14 individuals with pre-manifest and early stage HD. The intervention will entail one face-to-face coaching session (approximately 1 hour), and three remote video sessions (via secure Webex connection via computer or smart phone, or phone call if internet/smart phone is not available to participant) lasting approximately 20 minutes. Participants will also be given FitBit wearable activity monitors to allow for self- monitoring of physical activity for use during the 4-month intervention. Participants will be evaluated at baseline and again 4 months later on a range of exploratory outcomes including physical activity, self efficacy, disease-specific motor and cognitive function, walking endurance and strength. Results from this study will be used to make relevant adaptations to prepare for a multi-site randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* For premanifest - Confirmatory genetic testing for Huntington disease (HD) and diagnostic confidence score of 0-3 on Unified Huntington Disease Rating Scale, indicating pre-manifest disease state. For manifest HD - Confirmatory genetic testing for HD or confirmed clinical diagnosis of HD by neurologist
* Successful completion of Physical Activity Readiness Questionnaire (PAR-Q), or medical clearance from General Practioner
* For potential participants over age 60, a minimum score of 24 on the Mini-Mental State Examination (MMSE) (completed within 3 months) will be required for capacity to consent.
* For potential participants age 60-65, successful pass of electrocardiogram screen will be required.

Exclusion Criteria:

* Musculoskeletal injury that would interfere with participation in an exercise program
* Currently participating in a structured exercise program 3 times per week or more
* Uncontrolled psychiatric or behavioral problems that would interfere with participation in an exercise program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity (daily step counts) at 4 months | 4 months
  Physical activity as measured by waist worn device (Actigraph)

SECONDARY OUTCOMES:
Change in International Physical Activity Questionnaire (IPAQ) metabolic equivalent of task at 4 months | 4 months
  Questionnaire evaluating level of physical activity over past 7 days
Change in Lorig self efficacy scale at 4 months | 4 months
  Self efficacy questionnaire
Change in 6 minute walk distance at 4 months | 4 months
  Endurance measured by 6 minute walk test - distance completed over 6 minutes of walking
Change in grip strength at 4 months | 4 months
  Hand strength as measured with hand held dynamometer
Change in HD-PRO-TRIAD at 4 months | 4 months
  Questionnaire evaluating disease-specific measure of HD symptoms (cognitive, emotional and motor function)
Change in Unified Huntington Disease rating scale Total Motor Score at 4 months | 4 months
  Disease-specific measure of motor function
Change in Behavioral Regulation in Exercise Questionnaire (BREQ 2) at 4 months | 4 months
  A 19 item questionnaire measuring stages of self determination continuum
Change in Unified Huntington Disease Rating Scale Cognitive battery at 4 months | 4 months
  Disease-specific cognitive function as measured by Unified Huntington Disease Cognitive battery (Stroop, Symbol digit modality and verbal fluency)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University, New York, New York, United States